CLINICAL TRIAL: NCT00199511
Title: Comparison of Equiosmolar Doses of Mannitol 20% Versus Hypertonic Saline 7.5% Infusion in the Reduction of Brain Bulk During Elective Craniotomies for Supratentorial Brain Tumor Resection
Brief Title: Hypertonic Saline 75% vs Mannitol 20%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-05-154
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Brain Tumor; Tumor, Brain; Brain Neoplasm; Neoplasm, Supratentorial; Tumor, Supratentorial
Keywords: Brain Tumor; Intracranial Pressure; Osmolarity; Seric; Hypertonic Solution
MeSH Terms: conditions — Brain Neoplasms; Supratentorial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Administration of Hypertonic Solution 7.5% vs Mannitol 20%

SUMMARY:
The purpose of this study is to evaluate the effect of Hypertonic Saline 7.5% vs Mannitol 20% on brain bulk (using a 4 point scale), intracranial pressure (subdural catheter)and the changes on serum and urinary Na, K and Osmolarity during elective craniotomy for brain tumor resection.

DETAILED DESCRIPTION:
Raised intracranial pressure occurs following an expansion of an intracranial mass e.g. hematoma or brain tumor and if left untreated, can lead to brain ischemia, stroke and death.

Strategies for reducing raised intracranial pressure include hyperventilation, use of a hyperosmolar agent and the evacuation of the intracranial mass.

The two hypertonic solutions most commonly used are Mannitol 20% and Hypertonic Saline 7.5%.

During elective neurosurgical removal of a brain tumour, the anesthesiologist needs to reduce intracranial pressure and provide good operating brain conditions to avoid brain ischemia.

Currently, Mannitol 20% is routinely used intra-operatively in these patients to reduce brain bulk and intracranial pressure and to improve brain operating conditions.

However, Mannitol itself can cause secondary effects that can be deleterious to the neurological patient. Mannitol causes a diuresis which may lead to systemic hypovolemia and hypotension, and adverse changes in serum and urinary sodium, potassium and osmolarity.

Experience with Hypertonic saline 7.5%, has been mainly in brain injured patients either in the Emergency Dept or in the Intensive care setting. There is growing evidence that Hypertonic saline 7.5% is just as effective as Mannitol 20% in reducing raised intracranial pressure, especially in traumatic brain injury and it has become a widely accepted form of treatment. One of the advantages of Hypertonic saline is that it does not cause a diuresis and therefore less likely to cause hypotension and hypovolemia. While transient hypernatremia has been observed after the administration of hypertonic saline, there have been no clinical consequences.

Unfortunately there have been only two studies which compared the effectiveness of Hypertonic saline and Mannitol during elective brain surgery. One of them, Gemma et al, failed to demonstrate any difference in the reduction of brain bulk between Mannitol and Hypertonic saline. However the 2 solutions used had different osmolarities and this may have had a confounding effect on the results. In the other study (published in Polish), the authors found a 20% reduction in brain bulk in favour of hypertonic saline. In view of these two opposing findings, we feel that another investigation is warranted.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I - 3.
* Age >18 years.
* Scheduled for elective craniotomies for supratentorial brain tumour resection.
* Written informed consent.

Exclusion Criteria:

* Within the past six months, a history of unstable angina pectoris and/or having a myocardial infarction.
* Electrocardiogram abnormalities indicating severe ischemia.
* Congestive heart failure.
* Glasgow coma sore < 9
* Refusal to participate or refusal to agree to randomization.
* Known renal failure
* Known poorly controlled diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162
Dates: Start 2005-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Surgeon's assessment of brain bulk.
ICP reduction

SECONDARY OUTCOMES:
Changes in intracranial pressure
Changes in serum and urine levels of sodium, potassium and osmolarity.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary A Craen, MD, Principal Investigator — Associate Proffesor UWO
Locations (1):
- University Hospital LHSC, London, Ontario, Canada